CLINICAL TRIAL: NCT04590404
Title: Metabolism Informed Smoking Treatment in Medicaid and Medicare Patients: The MIST RCT
Brief Title: Metabolism Informed Smoking Treatment: The MIST RCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Hilary Tindle, Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 2046; 5R01CA232516-03 (NIH)
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Nicotine Replacement Therapy; Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIST (Metabolism-Informed Smoking Treatment) (Experimental): At hospital discharge, participants randomized to the MIST precision care arm will receive a prescription for medication (either varenicline or NRT). Post discharge, participants will receive automated phone calls via TelASK to promote continued engagement. Medication prescriptions will be informed by nicotine metabolism (i.e., NMR result) such that faster metabolizers are prescribed varenicline and slower metabolizers are prescribed NRT.
  Interventions: Behavioral: Post-discharge automated phone calls (IVR) with option to connect with a tobacco coach.; Drug: Nicotine Replacement Therapy; Drug: Varenicline; Other: Metabolism Informed Smoking Treatment (Nicotine metabolite ratio (NMR)-based selection of pharmacotherapy)
- Usual Care (Active Comparator): At hospital discharge, participants randomized to the Usual Care arm will receive a prescription for medication (either varenicline or NRT). Post discharge, participants will receive automated phone calls via TelASK to promote continued engagement. Medication prescription will not be informed by nicotine metabolism.
  Interventions: Behavioral: Post-discharge automated phone calls (IVR) with option to connect with a tobacco coach.; Drug: Nicotine Replacement Therapy; Drug: Varenicline

INTERVENTIONS:
Behavioral: Post-discharge automated phone calls (IVR) with option to connect with a tobacco coach. — Automated calls to assess smoking status, medication use, and additional support for quit attempt.
Drug: Nicotine Replacement Therapy — FDA-approved forms of nicotine replacement therapy for smoking cessation.
Drug: Varenicline — FDA-approved smoking cessation medication.
  Other Names: Chantix
Other: Metabolism Informed Smoking Treatment (Nicotine metabolite ratio (NMR)-based selection of pharmacotherapy) — Nicotine metabolite ratio (NMR)-based selection of pharmacotherapy. NMR is a blood test to measure how fast the body breaks down nicotine.
  Arms: MIST (Metabolism-Informed Smoking Treatment)

SUMMARY:
This phase 3 randomized controlled trial will test Metabolism-Informed Smoking Treatment (MIST), a precision approach to smoking treatment that biologically tailors medication selection to nicotine metabolism.

DETAILED DESCRIPTION:
This is a randomized controlled trial to compare effects of MIST versus usual care (UC) interventions on the outcomes below.

Objectives:

* Abstinence as defined by biochemically-verified self-reported 7-day point prevalence abstinence at 6 m (1° study outcome) and 12 m (2° outcome).
* Clinical practice implementation as measured by participant self-reported medication adherence at months 1 and 3, self-reported receipt of prescription for smoking cessation medication after hospital discharge, and whether the prescription was tailored to the NMR result.

Exploratory Objective:

- Longitudinal assessment of health care utilization visits (ER and hospitalization) for 12 months following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older
* be enrolled in an insurance plan that supports prescription coverage for smoking cessation medication (such as Medicare part D, Medicaid, or private insurance) to facilitate bedside delivery of medications prior to hospital discharge
* have a regular provider/PCP
* agree to quit or try to quit smoking upon hospital discharge
* be a daily smoker when smoking normally during the month prior to entering the hospital
* be medically eligible to use varenicline
* be medically eligible to use nicotine replacement therapy
* have received discharge medication recommendations from a tobacco counselor
* agree to take smoking cessation medication (i.e., varenicline OR nicotine replacement therapy) home and consider using it
* have a cell phone or landline that can be reached directly (i.e., without transfer)
* have a permanent address where they live and can receive mail
* estimated life expectancy of at least one year or greater

Exclusion Criteria:

* insufficient time to perform and complete the enrollment process
* barrier to effective communication (including low English proficiency)
* not cognitively able to participate in the study
* too ill, on hospice, or physically unable to participate in the follow-up process
* previously completed the MIST study or is currently enrolled in a quit smoking study that involves a medication-based treatment
* estimated life expectancy of less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Tindle, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center ViTAL, Vanderbilt Center for Tobacco, Addiction, and Lifestyle General Internal Medicine and Public Health 2525 West End Ave, Suite 450, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a tertiary care hospital in the US Mid-South from November 17, 2020 to September 29, 2023.
Pre-assignment Details: 5 participants were removed pre-randomization assignment by PI due to new information, discovered post-consent, indicating ineligibility.
Groups:
- MIST (Metabolism-Informed Smoking Treatment): All patients had a tobacco treatment consult and NMR measured by LC-tandem mass spectroscopy before randomization; all received 3 months of medication (varenicline or combination nicotine replacement therapy (NRT)) and access to tobacco counseling. The MIST intervention used NMR to select medication (Fast Metabolizers NMR≥0.31-varenicline; Slow Metabolizers NMR <0.31-NRT).
- Guideline-Based Care: All patients had a tobacco treatment consult and NMR measured by LC-tandem mass spectroscopy before randomization; all received 3 months of medication (varenicline or combination nicotine replacement therapy (NRT)) and access to tobacco counseling. Medication was selected by shared decision making. Guideline-based care participants were not informed of NMR results.
Period: Overall Study
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
Started | 294 | 307
1-month Survey | 259 | 271
3-month Survey | 246 | 264
6-month Survey | 247 | 261
12-month Survey | 235 | 246
Completed | 271 | 288
Not Completed | 23 | 19
Not completed — Death | 16 | 17
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care | Total
Number analyzed (Participants) | 294 | 307 | 601
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 231 | 220 | 451
  >=65 years | 63 | 87 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.88 (11.60) | 56.45 (11.53) | 56.17 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 136 | 263
  Male | 167 | 171 | 338
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 287 | 300 | 587
  Unknown or Not Reported | 2 | 3 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 58 | 66 | 124
  White | 224 | 239 | 463
  Unknown or Not Reported | 7 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 294 | 307 | 601

OUTCOME MEASURES:

1. Primary Outcome: Biochemically-validated Past 7-day Point Prevalence Tobacco Abstinence
Time Frame: 6 months
Population: Randomized participants were analyzed. Participants with missing self-report or biochemical verification data were assumed to be smoking (missing=smoking).
Measure: Count of Participants; unit: Participants
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
Number analyzed (Participants) | 294 | 307
Participants | 54 | 49
Statistical Analysis 1: Comparison: MIST (Metabolism-Informed Smoking Treatment) vs Guideline-Based Care; The primary outcome was biochemically-verified self-reported 7-day point prevalence abstinence (7dPPA) at 6 months. We modeled outcomes using logistic regression adjusted for randomization stratification factors and plan to quit (stay quit vs. try); Test type: Superiority; p = 0.461, Regression, Logistic; Adjusted for arm, randomization strata (cigarettes/day (CPD), insurance category, cardiac admission, NMR category), & plan to quit after discharge; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.76 to 1.82]

2. Secondary Outcome: Biochemically-validated Past 7-day Point Prevalence Tobacco Abstinence
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
Number analyzed (Participants) | 294 | 307
Participants | 49 | 51
Statistical Analysis 1: Comparison: MIST (Metabolism-Informed Smoking Treatment) vs Guideline-Based Care; The primary outcome was biochemically-verified self-reported 7-day point prevalence abstinence (7dPPA) at 12 months. We modeled outcomes using logistic regression adjusted for randomization stratification factors and plan to quit (stay quit vs. try); Test type: Superiority; p = 0.99, Regression, Logistic — Adjusted for arm, randomization strata (cigarettes/day (CPD), insurance category, cardiac admission, NMR category), & plan to quit after discharge; Odds Ratio (OR) = 1.0, 95% CI 2-sided [0.64 to 1.54]

3. Secondary Outcome: Self-reported Medication Adherence Over the Past 7 Days
Description: Participants taking any stop-smoking medications in past 7 days at 1 AND/OR 3 month surveys, also includes those who reported completing their course of medication at 3 months.
Time Frame: 1, 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
Number analyzed (Participants) | 294 | 307
Participants | 234 | 232

4. Secondary Outcome: Self-reported Receipt of Prescription for Smoking Cessation Medication Subsequent to the Initial Study Medication Prescription
Description: Randomized participants who reported having an office visit with PCP or regular healthcare provider and reported receiving a medication recommendation or prescription (since study enrollment; 1, 3, 6, or 12 months). Some participants may have reported receiving more than 1 prescription over the course of the 12 months.
Time Frame: Up to 12 months after hospital discharge
Population: Of note, 395 participants were missing for this measure due to report of not having an office visit and/or non-completion of all follow-up surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
Number analyzed (Participants) | 294 | 307
Participants | 70 | 74

ADVERSE EVENTS:
Time Frame: 12 months
Description: Other (non-serious) AEs are restricted to those that participants initially self-reported as "Severe" on follow-up surveys and were determined to be non-serious by PI review.
Arm/Group | MIST (Metabolism-Informed Smoking Treatment) | Guideline-Based Care
All-Cause Mortality (participants affected / at risk) | 16/294 | 17/307
Serious Adverse Events (participants affected / at risk) | 140/294 | 131/307
Other Adverse Events (participants affected / at risk) | 84/294 | 90/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MIST (Metabolism-Informed Smoking Treatment) (N=294) | Guideline-Based Care (N=307)
Anxiety (includes nervousness and panic attacks) (Psychiatric disorders) | 2 (2) | 6 (7)
Depressed mood (Psychiatric disorders) | 0 (0) | 7 (7)
Emergency Medical Visit (Cardiac disorders) | 9 (11) | 9 (10)
Emergency Medical Visit (Surgical and medical procedures) | 73 (159) | 76 (175)
Medication Side Effects (Product Issues) | 3 (3) | 0 (0)
Scheduled Medical Procedure (Cardiac disorders) | 5 (5) | 3 (3)
Scheduled Medical Procedure (Investigations) | 1 (1) | 0 (0)
Scheduled Medical Procedure (Surgical and medical procedures) | 26 (34) | 31 (36)
Hospital Admission (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hospital Admission (Cardiac disorders) | 16 (18) | 13 (15)
Hospital Admission (Endocrine disorders) | 0 (0) | 1 (1)
Hospital Admission (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hospital Admission (General disorders) | 0 (0) | 2 (2)
Hospital Admission (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hospital Admission (Infections and infestations) | 7 (8) | 5 (5)
Hospital Admission (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Hospital Admission (Investigations) | 0 (0) | 1 (1)
Hospital Admission (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Hospital Admission (Renal and urinary disorders) | 4 (8) | 8 (8)
Hospital Admission (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Hospital Admission (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hospital Admission (Surgical and medical procedures) | 26 (28) | 17 (19)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MIST (Metabolism-Informed Smoking Treatment) (N=294) | Guideline-Based Care (N=307)
Agitation and/or irritability (General disorders) | 12 | 18
Anxiety (includes nervousness and panic attacks) (Psychiatric disorders) | 15 | 21
Restlessness (General disorders) | 15 | 22
Headaches (Nervous system disorders) | 14 | 16
Fatigue (General disorders) | 19 | 30
Insomnia (General disorders) | 32 | 29

LIMITATIONS AND CAVEATS:
For context, this study began in 2020 at the start of the 2019 COVID pandemic, and was subject to delays associated with this global emergency. Additionally, in 2021 the study was impacted by the global recall of varenicline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT04590404/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04590404/ICF_001.pdf